CLINICAL TRIAL: NCT01083459
Title: Impact of PCV on Disease and Colonization Among Native American Communities
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Pfizer (Industry)
Responsible Party: Principal Investigator, Katherine O'Brien, Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: R01MD004011-01 (NIH)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Pneumococcal Nasopharyngeal Colonization; Invasive Pneumococcal Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCV13 immunized: Children who receive the 13-valent pneumococcal conjugate vaccine
- PCV13 unimmunized: PCV13 unimmunized Household members of PCV13 immunized children

SUMMARY:
The purpose of this study is to determine the impact of pneumococcal conjugate vaccine on carriage of pneumococcus in the nasopharynx and on the incidence of invasive pneumococcal disease in the community.

DETAILED DESCRIPTION:
Pneumococcus is a bacterium that healthy people commonly have in their nose and throat; this is called pneumococcal 'carriage'. Carriage is usually harmless, but can progress to serious disease like pneumonia, meningitis, and blood stream infections or to less serious, but burdensome, diseases like sinusitis or ear infections. Infants and the elderly bear the greatest burden of pneumococcal disease with over 800,000 annual global deaths from this germ among children under 5 years of age. Furthermore, pneumococcus has developed resistance to antibiotics making it increasingly difficult to treat pneumococcal infections. Within the United States some Native American groups, like the Navajo and the White Mountain Apache tribes, suffer from pneumococcal disease much more often than people in the general US population. We don't know why pneumococcus disproportionately afflicts these communities, but we know this health disparity can be significantly reduced through vaccination. In 2000, for the first time a pneumococcal vaccine designed specifically for infants, called PCV7, became available and was put into routine use among Navajo and Apache as well as the general US population. PCV7 contains the 7 most common of the >90 pneumococcal strains that exist. Although PCV7 is only given to infants and toddlers, it impacts pneumococcal disease throughout the community because it not only protects vaccinated infants from disease it also protects them against NP colonization. Infants and children are the main transmitters of pneumococcal colonization in the community so any change in their carriage affects the whole population of pneumococcal germs circulating within the family and community. Reductions in pneumococcal disease caused by the 7 types in PCV7 have exceeded expectations, especially among Navajo and Apache where we have seen virtually no cases in over 5 years. But, PCV7 has had the unintended consequence of increasing the amount of pneumococcal disease from some pneumococcal types that are not in PCV7. Therefore a new vaccine to protect against 13 pneumococcal strains, called PCV13, has been developed and is about to be licensed and used (expected licensure Q4/2009). This project aims to reveal the impact of PCV13 on pneumococcal disease and carriage of strains which move from person to person within the Navajo community. We specifically intend to find out if use of PCV13 has an effect on disease and carriage of the 6 additional strains in the vaccine and to find out if PCV13 will result in the emergence of new pneumococcal serotypes within the community, like PCV7 did. This information will allow us to design vaccine strategies to meet these new patterns of pneumococcal disease and stay at least one step ahead of the organism changes. It will also provide the evidence on which rational policies for PCV13 use among Navajo can be made. This has been essential information in past experiences of vaccine shortages, where Navajo communities were given priority for vaccine use. We also propose to explore the correlations between pneumococcal colonization and viral infection of the nasopharynx to establish if there is enhanced risk of pneumococcal colonization in the setting of viral co-infection and if that enhances the risk of developing disease. To achieve the overall objectives we propose pulling together three types of information (1) effect of PCV13 on nasopharyngeal colonization with pneumococcus and viral pathogens (2) effect of PCV13 on disease and (3) use of PCV13 in the community.

ELIGIBILITY:
Inclusion Criteria:

* American Indian children and their families (i.e. people of all ages) who live in the Whiteriver, Fort Defiance, Chinle, Gallup, Shiprock Service Units are eligible to participate in the carriage portion of the study.

Exclusion Criteria:

* Anyone with a congenital anomaly of the nasopharynx would not be eligible to participate in the carriage portion of the study

Min Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population for the nasopharyngeal study is American Indian children 7-24 months of age (index child) and their adult and child household members who reside in the Whiteriver, Shiprock, Chinle, Fort Defiance and Gallup service units on the White Mountain Apache and Navajo reservations. In addition those children and adults who have close contact with the index child but may not live in the same household as the child are eligible to participate. This may be relatives or close contacts of the index child who reside in the same family compound (a compound is a group of homes in close proximity to each other) but do not live in the same household as the index child.
Sampling Method: Non-Probability Sample
Enrollment: 6628 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Nasopharyngeal carriage or Invasive Pneumococcal Disease caused by a PCV13 serotype | Before PCV13 introduction and after 1 and 2 years of PCV13 use

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L O'Brien, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Lindsay R Grant, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - White Mountain Apache reservation, Whiteriver, Arizona
  - Navajo reservation, Gallup, New Mexico